CLINICAL TRIAL: NCT03352856
Title: Randomized, Double-blind, Placebo Controlled Food Challenge for the Assessment of Non-allergenicity of Refined Barley Starch in Cereal Allergic Patients
Brief Title: Food Challenge With Barley Starch as Active Comparator
Acronym: BALA
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: Lyckeby Starch AB (Industry)
Collaborators: FinnMedi Oy (Industry); Oy Medfiles Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MF20142700/BALA
Record Dates: First submitted 2017-10-02; First posted 2017-11-24 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2018-11

CONDITIONS: Allergy;Food; Allergy Wheat
Keywords: Cereal allergy; barley starch, DBPC
MeSH Terms: conditions — Food Hypersensitivity; Wheat Hypersensitivity | interventions — Starch

STUDY DESIGN:
Intervention Model Description: Double-blind, cross-over, randomly allocated, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Highly purified barley starch packed in sachets; Increasing doses given at clinic as follows: 0.6 g, 2 g, 6 g and 18 g. If required, continued at home with 2 x 18 g daily for 5 days.
  Interventions: Other: Barley starch
- Placebo (Placebo Comparator): Maize starch packed in sachets; Increasing doses given at clinic as follows: 0.6 g, 2 g, 6 g and 18 g. If required, continued at home with 2 x 18 g daily for 5 days.
  Interventions: Other: Maize starch

INTERVENTIONS:
Other: Barley starch — Highly purified barley starch
  Arms: Active
Other: Maize starch — Maize starch
  Arms: Placebo

SUMMARY:
Aim of the present study is to verify in a double-blind placebo controlled food challenge (DBPCFC) test that highly purified barley starch ingredient do not cause allergic reaction in subjects most potential to get allergic reaction due to ingredient. Hypothesis is that none of the cereal (mostly primarily wheat) allergic subject recruited to the study will obtain allergic reaction neither to placebo nor to the test ingredient. Scoring of symptoms during the challenges will be based on PRACTALL.

ELIGIBILITY:
Inclusion Criteria:

* Age = 1-20 years
* Diagnosed or suspected cereal allergy (at least to one of the following cereals wheat, barley or rye)
* Response to cereal proteins confirmed within 2 months in an oral food challenge (OFC)* OR response to cereal proteins confirmed in an OFC more than 2 months ago but clinically verifiable and documented ongoing cereal allergy at the time of inclusion OR diagnosis confirmed in an OFC with wheat performed as part of the study procedures.
* Voluntarily signed informed consent (including willingness to refrain from cereal containing foods for 1 week before intervention period and be exposed to cereal proteins in the test for eligibility)

Exclusion Criteria:

* Complex food allergy which make elimination diet impossible to accomplish
* Patients experiencing unstable or exacerbated atopic disease, such as asthma, atopic dermatitis (AD), urticaria, or allergic rhinitis.
* Diseases and conditions that might affect safety. Patients should not be challenged if they have chronic medical the event of anaphylaxis/treatment of anaphylaxis. Examples of such conditions include unstable angina pectoris, cardiac disease or dysrhythmias, severe chronic lung disease.
* Pregnancy should be ruled out by testing or based on history (e.g, before menarche) as appropriate
* Use of oral corticosteroids. Inhaled and topical steroids or anti-inflammatory medications, such as calcineurin inhibitors or leukotriene antagonists and b-agonists, used at the lowest doses possible and on an established schedule by using fixed doses of medication to maintain a low and stable baseline of atopic disease. Latter medication can usually be continued because their use is unlikely to significantly influence challenge outcomes and their withdrawal might result in exacerbations, affecting disease management and challenge interpretation.
* Use of antihistamines during the last 4 days before DBPC challenge or period of 5 half-lives of specific agent.
* Prolonged high dose steroids, omalizumab, or possibly other new drugs to control atopic disease upon decision of investigator.
* Aspirin/nonsteroidal anti-inflammatory drugs, angiotensin converting enzyme inhibitors, alcohol, antacids and β-blockers upon the decision of the investigator
* Any chronic condition or its medication that affect immune system

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-10-13 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Challenge outcome according to PRACTALL -score | 12-24 days (including 2 blinded challenges)
  Allergic reaction to active or placebo. Scoring and decision making based on PRACTALL as defined by Sampson et al., J Allergy Clin Immunol. 2012 Dec;130(6):1260-74.

SECONDARY OUTCOMES:
Severity of atopic dermatitis according to SCORAD-index | 12-24 days (including 2 blinded challenges)
  Worsening of atopic dermatitis
Symptom diary | 12-24 days (including 2 blinded challenges)
  Subjective symptoms based on diary

CONTACTS AND LOCATIONS:
Overall Officials: Marita Paassilta, MD, Docent, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No